CLINICAL TRIAL: NCT06283134
Title: A Clinical Study to Evaluate the Safety and Efficacy of Recombinant Human nsIL12 Oncolytic Adenovirus Injection (BioTTT001) in Combination With Toripalimab and Regorafenib in Patients With Liver Metastases From Colorectal Cancer
Brief Title: A Clinical Study of BioTTT001 in Combination With Toripalimab and Regorafenib in Patients With Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University, China (Other)
Collaborators: Beijing Bio-Targeting Therapeutics Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, Funan Liu, professor, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJCT-CMU1H-02
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Metastatic
Keywords: oncolytic virus; colorectal Cancer; liver metastasis; hepatic artery infusion
MeSH Terms: conditions — Colorectal Neoplasms | interventions — toripalimab; regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy with BioTTT001 hepatic artery infusion , Regorafenib and Toripalimab (Experimental): This study includes a dose escalation phase and a dose expansion phase. The dose escalation phase will adopt a 3+3 design. Subjects were first treated with BioTTT001 monotherapy (hepatic artery infusion, administered on D1 and D8 for a total of two doses) after enrollment. If the subject does not develop dose-limiting toxicity (DLT) in the monotherapy stage and is judged to be safe and tolerable by the investigator, the subject will enter the treatment phase of BioTTT001 in combination with toripalimab and regorafenib 2 weeks after the first dose of BioTTT001 ( toripalimab 160mg iv. D1 and D15 , BioTTT001 5×10^9 viral particle (VP)/5×10^10 VP/1×10^11 VP hepatic arterial infusion (HAI.) D2 and D16 , regorafenib 80 mg Po. D1-D21; 4 weeks per cycle). In the dose expansion phase, different dose groups can be expanded, and the total number of enrolled subjects is expected to be 23~48 for further safety, tolerability, pharmacokinetics and preliminary efficacy evaluation.
  Interventions: Biological: BioTTT001 hepatic artery infusion; Drug: toripalimab; Drug: regorafenib

INTERVENTIONS:
Biological: BioTTT001 hepatic artery infusion — BioTTT001 monotherapy period: BioTTT001 5×10^9 VP/5×10^10VP/1×10^11 VP hepatic artery infusion, administered on D1 and D8, for a total of two doses after enrollment.
  BioTTT001 in combination with toripalimab and regorafenib period: BioTTT001 5×10^9 VP/5×10^10VP/1×10^11 VP hepatic artery infusion, D2 and D16, 4 weeks per cycle.
Drug: toripalimab — BioTTT001 in combination with toripalimab and regorafenib period: toripalimab 160mg intravenous D1 and D15, 4 weeks per cycle.
Drug: regorafenib — BioTTT001 in combination with toripalimab and regorafenib period: regorafenib 80 mg oral administration, D1-D21, 4 weeks per cycle.

SUMMARY:
This is a phase I, open-label clinical study of BioTTT001 in combination with Toraplizumab and Regorafenib in patients with liver metastases from colorectal cancer.

DETAILED DESCRIPTION:
This study includes a dose escalation phase and a dose expansion phase. The dose escalation phase will adopt a 3+3 design. Subjects were first treated with BioTTT001 monotherapy (hepatic artery infusion, administered on D1 and D8 for a total of two doses) after enrollment. If the subject does not develop dose-limiting toxicity (DLT) in the monotherapy stage and is judged to be safe and tolerable by the investigator, the subject will enter the treatment phase of BioTTT001 in combination with toripalimab and regorafenib 2 weeks after the first dose of BioTTT001 ( toripalimab 160mg iv. D1 and D15 , BioTTT001 5×10^9 viral particle (VP)/5×10^10 VP/1×10^11 VP hepatic arterial infusion (HAI.) D2 and D16 , regorafenib 80 mg Po. D1-D21; 4 weeks per cycle). In the dose expansion phase, different dose groups can be expanded, and the total number of enrolled subjects is expected to be 23~48 for further safety, tolerability, pharmacokinetics and preliminary efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18 to 70 years old (including the threshold), no gender restrictions;
2. Patients with a definitive histopathological or cytological diagnosis of colorectal cancer with hepatic metastases who have received and failed at least second-line standard therapy in the past, or who have been assessed by the investigator to be unsuitable for standard therapy;
3. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1;
4. WBC≥3.0×10^9/L; ANC≥1.5×10^9/L (without cytokine therapy within one week before the screening ); Hb≥90g/L(without blood transfusion within one week before the screening);PLT≥90×10^9/L(without Platelet transfusion or thrombopoietin (TPO) within one week before the screening)；ALT and AST≤5×ULN；Cr≤1.5×ULN or CCr>50mL/min; TBIL≤1.5×ULN; APTT≤1.5×ULN and INR/PT≤1.5×ULN；
5. ECOG 0~2；
6. Expected survival ≥ 3 months;
7. Consent to contraception；
8. Understand and voluntarily sign a written ICF and be willing to comply with all trial requirements.

Exclusion Criteria:

1. Known allergy to the investigational drug or its components;
2. Previous treatment with other adenovirus drugs;
3. Patients with active autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, etc.), except type 1 diabetes, hypothyroidism that only needs hormone replacement therapy, and skin diseases that do not need systemic treatment (such as vitiligo, psoriasis or alopecia);
4. Received treatment with nitrosourea or mitomycin C within 6 weeks before the first dose of BioTTT001; received oral fluorouracil and small molecule targeted drug therapy within 2 weeks or 5 half-lives of the drug within 2 weeks before the first dose of BioTTT001; received traditional Chinese medicine therapy with anti-tumor indications within 2 weeks before the first dose of BioTTT001; received chemotherapy, radiotherapy, biological therapy other than the drugs mentioned above within 28 days before the first dose of BioTTT001；
5. Patients who have not recovered from the adverse reactions of previous treatments (the treatment-related toxicity ≤ grade 2, except for alopecia, pigmentation or other tolerable events judged by the investigator ).
6. History of other malignancies (except cured basal cell skin cancer, cervical carcinoma in situ, Papillary carcinoma of thyroid gland, low-risk GIST etc.) within 5 years before study drug administration;
7. Patients who have undergone any major surgery (except needle biopsy, etc.) or severe trauma within 4 weeks before the first dose of BioTTT001;
8. Patients who have been treated with high-dose systemic corticosteroids (prednisone > 10 mg/day or equivalent doses) or other immunosuppressants within 2 weeks before the first dose of BioTTT001;
9. NYHA≥grade 3; LVEF<50%; male QTc>450 mms, female QTc>470 mms;
10. Patients with active tuberculosis or drug-induced interstitial lung disease；
11. Patients with active infection requiring systemic anti-infective therapy;
12. In a state of immunosuppression, such as severe combined immunodeficiency disease or concurrent opportunistic infections;
13. HBsAg positive, and blood HBV DNA≥100 IU/mL; anti-HCV positive; HIV positive; active syphilis;
14. Patients with pleural effusion and ascites with clinical symptoms that require repeated drainage;
15. Patients with central nervous system metastases or meningeal metastases with clinical symptoms;
16. Patients with contraindications to hepatic arterial perfusion therapy;
17. Pregnant or lactating women;
18. Patients with prior organ transplants;
19. Other reasons judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From the enrollment to 28 days after the end-of-trial visit (i.e. end of treatment or early termination visit)
  The incidence and severity of all types of adverse events evaluated based on NCI-CTCAE V5.0 assessment.
MTD | 42 days within the first dose of BioTTT001 injection
  Maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Overall survival(OS) | Every 3 months until consent withdraw, death, withdrawal study, or loss of follow-up, up to 100 weeks
  The time from the start of treatment to death for any cause
Progression-free survival (PFS) | At C1D28 of the combination therapy phase for the first time, and then every 8 weeks until disease progression, consent withdraw, death or end of study during the combination therapy phase, up to 100 weeks.
  The time from the start of treatment to progress disease or death for any cause
Objective response rate (ORR) | Imaging will be performed at C1D28 of the combination therapy phase for the first time, and then every 8 weeks during the combination therapy phase.
  Objective response rate (ORR) as assessed by the investigators
Plasma adenovirus (ADV) copies | 8 days within the first BioTTT001 injection dose
  Pharmacokinetic Study (PK): Copies of ADV in plasma at various sampling points.
ADV copies in various sites | 8 days within the first BioTTT001 injection dose
  Viral Shedding Analysis: Copies of ADV in swabs of rectal swabs, throat swabs, and urine samples at various sampling points.
Serum IL-12 level | 8 days within the first BioTTT001 injection dose
  Expression levels of IL-12 at various sampling points in serum.
Serum neutralizing antibody level | 8 days within the first BioTTT001 injection dose
  Immunogenicity assessment through adenovirus neutralizing antibody detection.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenning Wang, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy; Funan Liu, MD, Principal Investigator — The First Affiliated Hospital of China Medical Univeristy